CLINICAL TRIAL: NCT05557058
Title: A Prospective, Randomized, Single-Center, Early Feasibility Clinical Study Designed to Evaluate the Safety and Effectiveness of the GORE Glaucoma Drainage Implant (GORE GDI) in Subjects With Primary Open-Angle Glaucoma Uncontrolled by Hypotensive Medications or for Which Conventional Incisional Glaucoma Surgery Would be More Likely to Fail Due to Scarring
Brief Title: GORE Glaucoma Drainage Implant Clinical Study Dominican Republic
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDI 21-03
Record Dates: First submitted 2022-09-20; First posted 2022-09-27 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Primary Open-angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gore GDI High Device Arm (Experimental): Implantation of the GORE GDI High Device Configuration
  Interventions: Device: Gore Glaucoma Device Implant (GORE GDI)
- Gore GDI Low Device Arm (Experimental): Implantation of the GORE GDI Low Device Configuration
  Interventions: Device: Gore Glaucoma Device Implant (GORE GDI)

INTERVENTIONS:
Device: Gore Glaucoma Device Implant (GORE GDI) — Unilateral implantation of one of two different configurations of the GORE GDI

SUMMARY:
The objective of this early feasibility clinical study is to evaluate the safety and effectiveness of the GORE Glaucoma Drainage Implant (2 configurations) in subjects with primary open-angle glaucoma that is uncontrolled by hypotensive medications or for which conventional incisional glaucoma surgery would be more likely to fail due to scarring.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age 18 to 85 years, inclusive at screening visit
* A diagnosis of primary open-angle glaucoma (Shaffer angle ≥ 3 as seen on gonioscopy) at screening visit
* Medicated intraocular pressure at screening visit and the mean medicated diurnal IOP at baseline visit ≥ 18 mmHg and ≤ 40 mmHg by Goldmann Applanation Tonometry

Exclusion Criteria:

* Expected inability to implant the study device in the superotemporal quadrant (e.g., a lack of freely mobile conjunctiva to cover the entire implanted device in the superotemporal quadrant)
* Diagnosis of any active ocular disease or disorder (other than glaucoma) that requires treatment, where the disease or treatment could be reasonably expected to affect the vision or IOP during the duration of the study
* Prior corneal transplant surgery (full or partial thickness transplants) or clinically significant corneal dystrophy, e.g., Fuchs' dystrophy (> 12 confluent guttae) in the study eye
* Concurrent cataract surgery or anticipated need for cataract surgery (i.e., clinically significant cataract) in the study eye during the 12 months following implantation
* BCDVA worse than 20/200 in the fellow (non-study) eye at the screening visit and BCDVA of the fellow eye cannot be worse than that of the study eye.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | 6 months
  The proportion of treated eyes with ≥ 20% decrease in mean diurnal IOP at 6 months while maintaining the same or fewer number of hypotensive medications as at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Batlle Pichardo, M.D., Principal Investigator — Laser Center
Locations (1):
- Laser Center, Santo Domingo, Dominican Republic